CLINICAL TRIAL: NCT06404983
Title: A Comparative Evaluation of Opioid Free Anaesthesia Technique Versus the Conventional Technique in Oncological Breast Surgery
Brief Title: Opioid-free Anaesthesia in Breast Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Agathi Karakosta, Assistant Professor of Anaesthesiology, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27
Record Dates: First submitted 2024-03-27; First posted 2024-05-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Anesthesia; Pain, Postoperative; Pain, Chronic; Opioid Free Anaesthesia; Cancer Recurrence
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Chronic Pain | interventions — Ketamine; Lidocaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Free Anaesthesia (OFA group) (Experimental): Patients are randomly allocated to receive non-opioid anaesthesia. Intraoperative analgesia will be achieved by continuous intravenous administration of a mixture of dexmedetomidine, ketamine, and lidocaine.
  Interventions: Other: Opioid Free Anaesthesia (OFA)
- Conventional general anaesthesia (CGA group) (Active Comparator): Patients are randomly allocated to receive conventional general anaesthesia with intraoperative use of opioids at the discretion of the attending anaesthesiologist.
  Interventions: Other: Conventional General Anaesthesia (CGA)

INTERVENTIONS:
Other: Opioid Free Anaesthesia (OFA) — Patients are allocated to receive non-opioid anaesthesia intraoperatively. Patients will receive a mixture of dexmedetomidine, ketamine and lidocaine for intraoperative analgesia.
  Other Names: N.O.A.M (non-opioid anaesthetic mixture: dexmedetomidine, ketamine and lidocaine)
  Arms: Opioid Free Anaesthesia (OFA group)
Other: Conventional General Anaesthesia (CGA) — Patients are allocated to receive conventional general anaesthesia intraoperatively with the use of fentanyl and morphine for intraoperative analgesia.
  Other Names: O.A.M. (Opioid Anaesthetic Mixtute: fentanyl, morphine)
  Arms: Conventional general anaesthesia (CGA group)

SUMMARY:
Background:

Various analgesic modalities are adopted for perioperative analgesia in breast cancer surgeries. Opioid-free and opioid-sparing techniques are gaining popularity due to the lack of opioid-dependent undesirable effects, including respiratory depression, urinary retention, nausea and vomiting, constipation, itching, opioid-induced hyperalgesia, tolerance, addiction, and immune system disorders.

The goal of this prospective randomized clinical trial is to investigate the impact of opioid-free anaesthesia (OFA) versus conventional general anaesthesia (CGA) on postoperative analgesic requirements after breast cancer surgery (lumpectomy/mastectomy, with or without axillary lymph node excision).

Secondary objectives include comparative perioperative evaluation of cognitive function and postoperative adverse events during the first 48 hours atfter surgery. Comparative evaluation of intraoperative haemodynamics and hospital length of stay are also secondary objectives, as well as the incidence of neuropathic pain assessed by validated questionnaires at 3 and 6 months postoperatively.

During the preoperative screening, body measurements, age, gender, ASA (American Society of Anesthesiologists) physical status classification, educational level (using a 6-level scale: elementary, middle school, high school, higher education, higher education, and postgraduate/doctoral degree), home medication, and comorbidities (using the Charlson Comorbidity Index) are recorded.

Intraoperatively, the duration of anaesthesia, duration of surgery, associated intraoperative data (e.g., haemodynamic instability, adverse effects associated with protocol-administered pharmaceutical agents, etc.), and medications administered (type and quantity) are recorded.

The investigators expect to recruit at least 100 participants per group.

DETAILED DESCRIPTION:
INTRODUCTION. Opioids are the mainstay for achieving analgesia in the perioperative setting. Standard anaesthetic practice in breast cancer surgery involves balanced general anaesthesia with the use of opioids intra- and postoperatively. Opioid-free anaesthesia (OFA) is a relatively recent anaesthetic proposal whereby no opioid is administered intraoperatively (systemically, in neuraxial or peripheral block or intra-cavity) and the use of opioids is avoided throughout the perioperative period.

Non-opioid anaesthesia appears to provide adequate postoperative analgesia while protecting the patient from the side effects of opioids, which include respiratory depression, opioid-induced hyperalgesia, postoperative nausea/vomiting, cognitive dysfunction, etc. Recently, concerns have arisen regarding delayed healing, immunosuppression, and worsening of oncological outcomes in cancer patients due to the systemic use of opioids.

Side effects of opioids include:

* Respiratory depression
* Muscle stiffness
* Weakness of pharyngeal muscles
* Upper airway obstruction (muscle atony)
* Negative inotropic action
* Nausea, vomiting
* Ileus, constipation
* Urinary retention
* Tolerance and addiction
* Dizziness
* Excessive drowsiness and sleep disorder

BACKGROUND. During the past decade there has been a growing interest in opioid sparing and opioid free techniques for general anaesthesia. The international literature started to be enriched with interesting cases and small prospective studies supporting the benefits of this technique, especially in patients with morbid obesity. According to its proponents, this technique is characterized by: 1) sympatholysis, analgesia, and anaesthesia (MAC reduction) using dexmedetomidine, 2) analgesia with low-dose of ketamine, 3) administration of lidocaine adjunctively for anaesthesia and sympatholysis, 4) deep neuromuscular blockade until the end of the procedure, 5) use of sevoflurane or desflurane 0.7 to 1 MAC in O2/air and titration based on entropy or BIS monitoring and 6) administration of magnesium adjunctively for analgesia. Inadequate sympatholysis is corrected by titrated doses of clonidine, whereas excessive sympatholysis is treated by the administration of vasoconstrictors, preferably ephedrine because of its chronotropic action. In addition, dexamethasone, high-dose paracetamol, NSAIDs, and gabapentin can be used adjunctively in the context of multimodal management of surgical pain.

However, the OFA method is not without its disadvantages, of which the clinician should be aware. Ketamine can disrupt electrocerebral monitoring (e.g., BIS) for possible intraoperative vigilance, although according to the proponents of the method, intraoperative vigilance is only a possibility in incorrect use of the technique, and they argue that it is unlikely to occur if BIS is maintained below 60. The need for hemodynamic support with vasoconstrictor administration is an additional disadvantage, and there may be a need to infringe the OFA protocol to achieve ideal intubation conditions using small doses of short-acting opioids during induction of anesthesia. Also, a significant degree of cutaneous vasoconstriction may be observed, an expected a2 action of concern to the clinician. Finally, training of the nursing staff and familiarity with the method is required.

Despite the above disadvantages of the method, OFA is becoming increasingly popular because of its excellent management of postoperative pain, protecting the patient from surgical and opioid-induced hyperalgesia, and because of the minimization of the risk of respiratory depression in high-risk patients (COPD, sleep apnea, morbid obesity, etc.).

The prevalence of chronic postoperative pain after breast cancer surgery (mastectomy, lumpectomy, with or without lymph node excision) is high and according to recent reports is 29.8%. The OFA technique has been studied in breast cancer surgery. However, these are mostly small studies examining the efficacy of this technique in acute postoperative pain. The effect of the OFA technique on chronic pain after breast cancer surgery has not been studied so far.

GOAL OF STUDY. The primary objective of the study is to evaluate postoperative analgesia for breast cancer surgery of low and intermediate severity (mastectomy, lumpectomy, with or without lymph node excision). Specifically, this is a prospective comparative study of pain intensity and total postoperative consumption of opioids and other analgesics in patients who received general anesthesia under OFA protocol (OFA group) versus those who received general anesthesia using opioids (CGA group, conventional General Anaesthesia).

Secondary objectives are the evaluation of intraoperative haemodynamic stability by recording the total use of vasoactive substances, time of extubation, length of stay in the Post-Anesthesia Care Unit (PACU), and total length of hospitalization per study group. In addition, secondary objectives include the comparative recording of serious postoperative anaesthesia-related adverse events (postoperative hypoxaemia, postoperative ileus, nausea/vomiting, etc.) and the comparative study of cognitive function in the perioperative period.

As part of the second part of the study, all participants will be monitored for the development of postoperative chronic pain using specific tools. Chronic postsurgical pain assessment will be performed at 3 and 6 months postoperatively.

METHOD. The anaesthetic technique of the OFA group is based on the protocol of Mulier et al. The intraoperative management of the CGA group will follow standard clinical protocols. All patients will give written informed consent to be included in the study.

During the preoperative screening, somatometrics, age, gender, ASA (American Society of Anesthesiologists) physical status classification, educational level (using a 6-level scale: elementary, middle school, high school, higher education, higher education, and postgraduate/doctoral degree), home medication, and comorbidities (using the Charlson Comorbidity Index) are recorded.

Intraoperatively, the duration of anaesthesia, duration of surgery, and associated intraoperative data (e.g., haemodynamic instability, adverse effects associated with protocol-administered pharmaceutical agents, etc.) and medications administered (type and quantity) are being recorded.

The length of stay in the Post Anaesthesia Care Unit (PACU) and the length of stay in the hospital shall also be recorded. Serious adverse events related to general anaesthesia for 48 hours post-operatively shall be recorded.

The intensity of acute postoperative pain shall be assessed using the NRS (Numerical Rating Scale) scale (Numerical Rating Scale, 0-10) at predefined intervals up to 48 hours postoperatively.

Participants' cognitive status, chronic postoperative pain, depression, anxiety, stress, and satisfaction will be assessed using validated questionnaires at 3 and 6 months after surgery.

STATISTICAL ANALYSIS. This is a prospective single-blind randomized clinical trial. Randomization will be carried out using sealed envelopes sorted based on computer-generated random numbers (Random Allocation Software).

Sample size calculation is based on a pilot study of 20 consecutive participants that was carried out in the University Hospital of Ioannina, with the primary outcome beeing the difference in NRS between groups at 1, 6, and 12 hours postoperatively, both at rest and at a deep breath.

Participant recruitment is expected to take up to 2 years, and the investigators expect to enroll at least 100 patients per study group.

Data analysis will be performed using Stata™ software (Version 10.1 MP, Stata Corporation, College Station, TX 77845, USA).

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* breast cancer surgery (mastectomy, lumpectomy, with or without lymph node excision) under general anaesthesia

Exclusion Criteria:

* under 18 years
* patient refusal
* opioid use (systemic or not) for any reason (e.g., chronic malignant pain)
* language barrier (difficulty in communicating in Greek language)
* allergy to the administered agents
* severe arrhythmia or other serious cardiac disease
* severe liver and kidney failure
* dementia, psychiatric diseases, and/or preoperative cognitive impairment

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-09-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia. | From PACU (Post Anaesthesia Care Unit) admission to 48 hours postoperatively.
  Postoperative level of analgesia assessed by the NRS (Numerical Rating Scale, ranging from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable).
Postoperative consumption of opioids. | From PACU (Post Anaesthesia Care Unit) admission to 48 hours postoperatively.
  Total postoperative consumption of opioids.

SECONDARY OUTCOMES:
Perioperative blood pressure measurements. | From the beginning of surgery to PACU (Post Anaesthesia Care Unit) discharge, assessed up to 48 hours.
  Intermittent blood pressure measurements (every 5 minutes) - blood pressure measured in mmHg.
Perioparative pulse measurements. | From the beginning of surgery to PACU (Post Anaesthesia Care Unit) discharge, assessed up to 48 hours.
  Intermittent arterial pulse measurements (every 5 minutes) - measured in beats per minute.
Perioperative consumption of ephedrine. | From the beginning of surgery to PACU (Post Anaesthesia Care Unit) discharge, assessed up to 48 hours.
  Total intravenous consumption of ephedrine, measured in milligrams.
Perioperative consumption of atropine. | From the beginning of surgery to PACU (Post Anaesthesia Care Unit) discharge, assessed up to 48 hours.
  Total intravenous consumption of atropine, measured in milligrams.
Perioperative consumption of phenylephrine. | From the beginning of surgery to PACU (Post Anaesthesia Care Unit) discharge, assessed up to 48 hours.
  Total intravenous consumption of phenylephrine, measured in milligrams.
PACU (Post Anaesthesia Care Unit) length of stay. | From the beginning of surgery to PACU (Post Anaesthesia Care Unit) discharge, assessed up to 48 hours.
  Minutes from PACU (Post Anaesthesia Care Unit) admission to PACU discharge.
Duration from end of anaesthesia to extubation. | From end of anaesthesia, defined by anaesthetic drug discontinuation, to removal of endotracheal tube, assessed up to 48 hours.
  Minutes from anaesthetic drug discontinuation to removal of endotracheal tube from the patient.
Postoperative episodes of nausea and/or vomiting. | From PACU (Post Anaesthesia Care Unit) admission to 48 hours postoperatively.
  Number of participants with postoperative recording of episodes of nausea/vomiting.
Postoperative pruritus. | From PACU (Post Anaesthesia Care Unit) admission to 48 hours postoperatively.
  Number of participants with postoperative recording of pruritus.
Postoperative paralytic ileus. | From PACU (Post Anaesthesia Care Unit) admission to 48 hours postoperatively.
  Number of participants with postoperative clinical signs of paralytic ileus.
Postoperative respiratory depression. | From PACU (Post Anaesthesia Care Unit) admission to 48 hours postoperatively.
  Number of participants with postoperative recording of hypoxaemic episodes (SpO2<90% with FiO2 (fraction of inspired oxygen) 21%)
Postoperative sedation. | From PACU (Post Anaesthesia Care Unit) admission to 48 hours postoperatively.
  Number of participants with postoperative sedation measured with the Ramsay Sedation Scale (ranging from +4 (a violent dangerous patient) to -5 (an unarousable patient)).
Postoperative headache. | From PACU (Post Anaesthesia Care Unit) admission to 48 hours postoperatively.
  Number of participants with postoperative episodes of headache, as assessed in a 4 rating scale (0: no headache to 3: severe headache).
Postoperative neuropathic pain assessed by the S-LANSS pain score. | From hospital discharge until 6 months postoperatively.
  Number of participants with postoperative neuropathic pain assessed by the use of the S-LANSS pain score (ranging from 0 to 24 points, where ≥12 points suggest the presence of neuropathic pain symptomatology).
Postoperative neuropathic pain assessed by the McGill questionnaire. | From hospital discharge until 6 months postoperatively.
  Number of participants with postoperative neuropathic pain assessed by the use of the McGill questionnaire (The present pain intensity (PPI) is based on a scale of 0-5, with 0 meaning no pain).
Postoperative depression and anxiety. | From hospital discharge until 6 months postoperatively.
  Number of participants with postoperative depression and anxiety assessed by the use of DASS21 tool, which is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress (the greater the score the greater the risk for depression, anxiety and stress).
Postoperative cancer recurrence. | From hospital discharge to 5 years postoperatively.
  Number of participants with postoperative cancer recurrence as assessed by examination of patient records (clinical examination, imaging testing, laboratory testing and biopsies that are part of the patient's follow-up protocol).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication and for a year afterwards.

REFERENCES:
- [Background] Wang K, Yee C, Tam S, Drost L, Chan S, Zaki P, Rico V, Ariello K, Dasios M, Lam H, DeAngelis C, Chow E. Prevalence of pain in patients with breast cancer post-treatment: A systematic review. Breast. 2018 Dec;42:113-127. doi: 10.1016/j.breast.2018.08.105. Epub 2018 Sep 4. PMID 30243159
- See also: Opioid free anaesthesia (OFA) a Paradigm shift? (Mulier JP) — http://www.researchgate.net/publication/278307444